CLINICAL TRIAL: NCT02909231
Title: One-year Patient Reported Outcomes Following Hospitalization for Trauma
Status: Terminated | Type: Observational
Why Stopped: Failed to recruit sufficient subjects
Sponsor: University of Calgary (Other)
Collaborators: Vancouver Coastal Health (Other Government); University of British Columbia (Other)
Responsible Party: Principal Investigator, Chris Grant, MD, Clinical Assistant Professor, University of Calgary
Other Study IDs: REB15-1860
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Wounds and Injuries
Keywords: Patient Outcome Assessment
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Foothills Medical Centre: Patients admitted to the Foothills Medical Centre trauma service (Calgary, AB) over four months.
- Vancouver General Hospital: Patients admitted to the Vancouver General Hospital trauma service (Vancouver, BC) over four months.

SUMMARY:
This study evaluates the three, six, and twelve month patient reported outcomes of people admitted two trauma centres in western Canada over a four month period. Participants are evaluated using the Trauma Outcome Profile and a custom survey instrument.

DETAILED DESCRIPTION:
This study intends to assess patient reported outcomes following discharge from trauma services at the Foothills Medical Centre (FMC) and Vancouver General Hospital (VGH). The investigators will survey participants with pen-and-paper surveys at three, six and twelve months following discharge from hospital. The survey instrument being used is the Trauma Outcomes Profile, which has been previously validated in this population, supplemented by a supplemental survey to help further describe resources this population has access to in their recovery. The results of these surveys will be compared with pre-injury health status, injury types, mechanisms, and discharge medications and treatments. The investigators anticipate enrolling 500 participants starting in October 2016. At the conclusion of the study the investigators will have a better understanding of patient reported functional outcomes after trauma and will be better positioned to design trauma rehabilitation systems to service this population.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the trauma service at VGH or FMC
* Age 18 or older
* resident of Canada

Exclusion Criteria:

* English language literacy
* Impairments in cognition, motor, or communication that limit the ability to complete a paper-based survey
* No fixed address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults admitted to the trauma service at either of the two level I trauma centres in Western Canada (Vancouver General Hospital, Vancouver, BC and Foothills Medical Centre, Calgary, AB) over a four month period.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Medium-term health-related quality of life | Up to one year
  Assessment at 3, 6 and 12 months using the Trauma Outcomes Profile survey instrument.

SECONDARY OUTCOMES:
Local resource use for trauma patients admitted to hospital | Up to one year
  Assessment at 3, 6, and 12 months using a custom survey to assess local resource use and perceived needs

CONTACTS AND LOCATIONS:
Overall Officials: Chris Grant, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No